CLINICAL TRIAL: NCT02293616
Title: Strength Testing After Nitrate Delivery (STAND) in ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00030880
Record Dates: First submitted 2014-11-13; First posted 2014-11-18 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Respiratory Failure
Keywords: ICU; Respiratory Failure; Weakness; Nitrate supplementation
MeSH Terms: conditions — Respiratory Insufficiency; Asthenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate Rich (Experimental): A nitrate rich beetroot juice supplement (Beet It Shot®, James White Drinks, UK) high in nitrates will be provided to the subjects. Subject's diet will be supplemented once daily while hospitalized up to 14 days with one 70 ml bottle containing 300 mg of dietary nitrate.
  Interventions: Dietary Supplement: Nitrate Rich Beetroot Juice
- Nitrate Depleted (Placebo Comparator): This group will consume a beetroot juice supplement (Beet It Shot®, James White Drinks, UK) that has had the nitrate removed from the beverage by the manufacturer. Patient's diet will be supplemented once daily with one 70 ml bottle while hospitalized up to 14 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nitrate Rich Beetroot Juice — Nitrate rich beetroot juice diet supplement will be consumed by subjects.
  Other Names: Beet It Shot®
  Arms: Nitrate Rich
Dietary Supplement: Placebo
  Arms: Nitrate Depleted

SUMMARY:
It is well documented that intensive care unit (ICU) patients have lower levels of skeletal muscle strength compared to non-ICU patients upon hospital discharge, and this weakness affects the patient's ability to perform basic activities of daily living upon hospital discharge and for extended periods thereafter. Recently, critically ill ICU patients have been shown to have lower nitric oxide levels. These patients often suffer from a disturbed homeostasis with circulatory and metabolic abnormalities that may potentially contribute to their ICU acquired weakness. Given the recent research showing dietary nitrate supplementation can increase nitric oxide levels and improve exercise tolerance in healthy and diseased older individuals, our aim is to investigate the importance of nitrate supplementation in ICU patients with focus on physical function and ICU acquired muscle weakness.

DETAILED DESCRIPTION:
The proposed study is an investigator initiated, double blind, placebo controlled experimental study designed to evaluate the effect of chronic NO3- supplementation via beetroot juice ingestion on the skeletal muscle strength and physical function in ICU patients. Patients will be randomized to receive either nitrate rich or nitrate depleted beetroot juice once daily during their ICU and hospital stay. Physical function and skeletal muscle strength will be measured at ICU (± 2 days) and hospital (± 2 days) discharge and 2 months (± 2 weeks) after enrollment. Plasma levels of nitrate and nitrite will be measured 1, 3 and 5 days after randomization into the trial and at ICU and hospital discharge. Skeletal muscle ultrasound will be performed to examine the size and echogenicity of patient muscles. Self-reported physical function will be measured using the Functional Performance Inventory Short Form (FPI-SF). The FPI-SF provides an overall score of patient self-reported functional performance in the areas of household maintenance, movement, family and social activities, work, avocation and recreation

ELIGIBILITY:
Inclusion Criteria:

* Age > 55 years
* Mechanically ventilated via an endotracheal tube or mask who have begun spontaneous breathing trials or extubated within the previous 24 hours
* Lung Injury as defined by a PaO2 / FiO2 < 300

Exclusion Criteria:

* Inability to walk without assistance prior to acute ICU illness (use of a cane or walkers not exclusions)
* Cognitive impairment prior to acute ICU illness (non-verbal)
* Acute stroke
* Body mass index (BMI) >50
* Neuromuscular disease that could impair weaning (myasthenia gravis, ALS, Guillain-Barre)
* Hip fracture, unstable cervical spine or pathological fracture
* Mechanically Ventilated > 80 hours
* Current hospitalization or transferring hospital stay > 7 days
* DNR/DNI on admission
* Cancer treatment within the last 6 months
* Moribund
* Participation in another research study
* On nitroglycerine or nitrate preparations used with angina or phosphodiesterase type 5 inhibitors
* Body mass less than 60 kg

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
physical function assessed using the Short Physical Performance Battery (SPPB) | 2 months
  The SPPB is based on timed measures of standing balance, walking speed, and ability to rise from a chair. Each performance measure is assigned a score ranging from 0 to 4, with 4 indicating the highest level of performance and 0 inability to complete the test. A summary score (range 0-12) will be calculated by adding the three scores.

SECONDARY OUTCOMES:
Plasma Nitrate and Nitrite Levels | 5 days
  Blood samples will be collected in 4 mL lithium heparin vials. Nitrate and nitrite will be measured separately using the ENO-20 NOx analyzer.
Skeletal muscle strength | 2 months
  Skeletal muscle strength will be measured in both upper and lower extremities. Hand grip strength in both hands will be measured using a hand held grip strength dynamometer. Additionally, an electronic strength dynamometer will be used to collect strength measures of the elbow flexion, elbow extension, shoulder flexion in the scaption plane, ankle dorsiflexion, knee extension and hip extension, bilaterally. Skeletal muscle ultrasound will be performed on upper and lower extremities bilaterally.
Hospital Length of Stay | 2 weeks
  The hospital calendar days (or any portion of a calendar day) at the enrolling hospital and at any long term acute care facility to which the subject is directly transferred.

CONTACTS AND LOCATIONS:
Overall Officials: D. Clark Files, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berry MJ, Morris PE. Early exercise rehabilitation of muscle weakness in acute respiratory failure patients. Exerc Sport Sci Rev. 2013 Oct;41(4):208-15. doi: 10.1097/JES.0b013e3182a4e67c. PMID 23873130
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Background] Fletcher SN, Kennedy DD, Ghosh IR, Misra VP, Kiff K, Coakley JH, Hinds CJ. Persistent neuromuscular and neurophysiologic abnormalities in long-term survivors of prolonged critical illness. Crit Care Med. 2003 Apr;31(4):1012-6. doi: 10.1097/01.CCM.0000053651.38421.D9. PMID 12682465
- [Background] Garland A, Dawson NV, Altmann I, Thomas CL, Phillips RS, Tsevat J, Desbiens NA, Bellamy PE, Knaus WA, Connors AF Jr; SUPPORT Investigators. Outcomes up to 5 years after severe, acute respiratory failure. Chest. 2004 Dec;126(6):1897-904. doi: 10.1378/chest.126.6.1897. PMID 15596690
- [Background] Groll DL, To T, Bombardier C, Wright JG. The development of a comorbidity index with physical function as the outcome. J Clin Epidemiol. 2005 Jun;58(6):595-602. doi: 10.1016/j.jclinepi.2004.10.018. PMID 15878473
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Kelly J, Fulford J, Vanhatalo A, Blackwell JR, French O, Bailey SJ, Gilchrist M, Winyard PG, Jones AM. Effects of short-term dietary nitrate supplementation on blood pressure, O2 uptake kinetics, and muscle and cognitive function in older adults. Am J Physiol Regul Integr Comp Physiol. 2013 Jan 15;304(2):R73-83. doi: 10.1152/ajpregu.00406.2012. Epub 2012 Nov 21. PMID 23174856
- [Background] Kenjale AA, Ham KL, Stabler T, Robbins JL, Johnson JL, Vanbruggen M, Privette G, Yim E, Kraus WE, Allen JD. Dietary nitrate supplementation enhances exercise performance in peripheral arterial disease. J Appl Physiol (1985). 2011 Jun;110(6):1582-91. doi: 10.1152/japplphysiol.00071.2011. Epub 2011 Mar 31. PMID 21454745
- [Background] Leidy NK. Psychometric properties of the functional performance inventory in patients with chronic obstructive pulmonary disease. Nurs Res. 1999 Jan-Feb;48(1):20-8. doi: 10.1097/00006199-199901000-00004. PMID 10029398
- [Background] Luiking YC, Deutz NE. Exogenous arginine in sepsis. Crit Care Med. 2007 Sep;35(9 Suppl):S557-63. doi: 10.1097/01.CCM.0000279191.44730.A2. PMID 17713409
- [Background] Lundberg JO, Weitzberg E, Gladwin MT. The nitrate-nitrite-nitric oxide pathway in physiology and therapeutics. Nat Rev Drug Discov. 2008 Feb;7(2):156-67. doi: 10.1038/nrd2466. PMID 18167491
- [Background] Mensinga TT, Speijers GJ, Meulenbelt J. Health implications of exposure to environmental nitrogenous compounds. Toxicol Rev. 2003;22(1):41-51. doi: 10.2165/00139709-200322010-00005. PMID 14579546
- [Background] Zimmerman JE, Kramer AA, McNair DS, Malila FM, Shaffer VL. Intensive care unit length of stay: Benchmarking based on Acute Physiology and Chronic Health Evaluation (APACHE) IV. Crit Care Med. 2006 Oct;34(10):2517-29. doi: 10.1097/01.CCM.0000240233.01711.D9. PMID 16932234
- [Derived] Gandotra S, Files DC, Shields KL, Berry M, Bakhru RN. Activity Levels in Survivors of the Intensive Care Unit. Phys Ther. 2021 Sep 1;101(9):pzab135. doi: 10.1093/ptj/pzab135. PMID 34097055